CLINICAL TRIAL: NCT00030914
Title: Phase III Comparison of Depomedroxyprogesterone Acetate (DPROV) to Venlafaxine for Managing Hot Flashes
Brief Title: Medroxyprogesterone Compared With Venlafaxine in Treating Hot Flashes in Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: NCCTG-N99C7; CDR0000069217 (Registry Identifier: PDQ (Physician Data Query)); NCI-P02-0204
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Hot Flashes
Keywords: hot flashes
MeSH Terms: conditions — Hot Flashes | interventions — Medroxyprogesterone; Venlafaxine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I: venlafaxine (Experimental): All patients complete a daily questionnaire regarding number of hot flashes beginning on day 1 and continuing for 7 weeks. Patients receive oral venlafaxine once daily for 6 weeks beginning on day 8. After week 7, patients with satisfactory efficacy may continue venlafaxine for up to 6 months. Patients with unsatisfactory efficacy may cross over to arm III.
  Patients are followed at months 2, 3, 4, 5, 6, 8, 10, and 12.
  Interventions: Drug: venlafaxine
- Arm II: medroxyprogesterone - long term (Experimental): All patients complete a daily questionnaire regarding number of hot flashes beginning on day 1 and continuing for 7 weeks. Patients receive medroxyprogesterone intramuscularly (IM) on days 8, 22, and 36 for a total of 3 injections. After week 7, patients with unsatisfactory efficacy may cross over to arm I.
  Patients are followed at months 2, 3, 4, 5, 6, 8, 10, and 12.
  Interventions: Drug: medroxyprogesterone
- Arm III: medroxyprogesterone - short term (Experimental): All patients complete a daily questionnaire regarding number of hot flashes beginning on day 1 and continuing for 7 weeks. Patients receive medroxyprogesterone IM once on day 8. After week 7, patients with unsatisfactory efficacy may cross over to arm I.
  Patients are followed at months 2, 3, 4, 5, 6, 8, 10, and 12.
  Interventions: Drug: medroxyprogesterone

INTERVENTIONS:
Drug: medroxyprogesterone
  Arms: Arm II: medroxyprogesterone - long term; Arm III: medroxyprogesterone - short term
Drug: venlafaxine
  Arms: Arm I: venlafaxine

SUMMARY:
RATIONALE: Medroxyprogesterone and venlafaxine may be effective in relieving hot flashes. It is not yet known whether venlafaxine is more effective than medroxyprogesterone in relieving hot flashes.

PURPOSE: Randomized phase III trial to compare the effectiveness of medroxyprogesterone with that of venlafaxine in treating women who are experiencing hot flashes.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of medroxyprogesterone administered as 1 injection vs medroxyprogesterone administered as 3 injections (closed to accrual as of 1/22/03) vs venlafaxine for hot flash alleviation in women with symptomatic hot flashes.
* Compare the toxic effects of these regimens in these patients.
* Determine whether there is cross resistance between these 2 drugs in these patients.
* Compare the 1-year efficacy of these regimens in these patients.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to age (18 to 49 vs 50 and over), current tamoxifen use (yes vs no), current raloxifene use (yes vs no), duration of hot flash symptoms (less than 9 months vs 9 months or more), and average frequency of hot flashes per day (2-3 vs 4-9 vs 10 or more). Patients are randomized to 1 of 2 treatment arms. (Arm II closed to accrual as of 1/22/03.)

All patients complete a daily questionnaire regarding number of hot flashes beginning on day 1 and continuing for 7 weeks. Patients are randomized to one of three treatment arms.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* History of breast cancer, ductal carcinoma in situ, or lobular carcinoma in situ (currently without evidence of malignant disease) OR
* Concerns about taking estrogen for fear of breast cancer
* Bothersome hot flashes, defined as occurrence at least 14 times per week and of sufficient severity as to make patient desire therapeutic intervention
* Presence of hot flashes for at least 1 month
* Hormone receptor status:

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Performance status:

* ECOG 0-1

Life expectancy:

* At least 6 months

Cardiovascular:

* No prior thromboembolic disease
* No uncontrolled hypertension (persistent diastolic blood pressure greater than 95 mm Hg and/or systolic blood pressure greater than 160 mm Hg)

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Chemotherapy:

* More than 4 weeks since prior antineoplastic chemotherapy
* No concurrent antineoplastic chemotherapy unless clinically appropriate

Endocrine therapy:

* More than 4 weeks since prior androgen or estrogen therapy
* More than 3 months since prior progesterone as part of hormone replacement therapy
* At least 1 year since any other progesterone therapy (including megestrol)
* No concurrent androgen, estrogen, or progestational agents unless clinically appropriate
* Concurrent tamoxifen, raloxifene, or aromatase inhibitors are allowed if started more than 4 weeks ago and continuation for more than 5 weeks is planned

Other:

* More than 2 weeks since prior agents for treatment of hot flashes (e.g., clonidine, Bellergal-S, or vitamin E of more than 400 mg per day)
* More than 1 year since prior antidepressants (including Hypericum perforatum [St John's Wort])
* No other concurrent antidepressants or monoamine oxidase inhibitors
* No other concurrent agents for treatment of hot flashes (e.g. clonidine, Bellergal-S, or vitamin E of more than 400 mg per day)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2002-04; Primary Completion 2006-02 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Compare the efficacy of the three regimens | Up to one year post-treatment

SECONDARY OUTCOMES:
Determine whether there is cross resistance between these 2 drugs in these patients | Up to 1 year post-treatment
Compare the 1-year efficacy of these regimens in these patients | Up to 1 year post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Charles L. Loprinzi, MD, Study Chair — Mayo Clinic
Locations (22):
- United States (22):
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin

REFERENCES:
- [Result] Loprinzi CL, Levitt R, Barton D, Sloan JA, Dakhil SR, Nikcevich DA, Bearden JD 3rd, Mailliard JA, Tschetter LK, Fitch TR, Kugler JW. Phase III comparison of depomedroxyprogesterone acetate to venlafaxine for managing hot flashes: North Central Cancer Treatment Group Trial N99C7. J Clin Oncol. 2006 Mar 20;24(9):1409-14. doi: 10.1200/JCO.2005.04.7324. Epub 2006 Feb 27. PMID 16505409